CLINICAL TRIAL: NCT02691299
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase III Clinical Trial in Patients With Advanced Non-squamous Non-small Cell Lung Cancer Treated With Fruquintinib
Brief Title: A Phase III Clinical Trial of Fruquintinib in Patients With Advanced Non-small Cell Lung Cancer
Acronym: FALUCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-013-00CH1
Record Dates: First submitted 2016-02-18; First posted 2016-02-25 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: NSCLC
Keywords: NSCLC
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (Active Comparator): All subjects will receive study treatment in 4-week cycles: Fruquintinib, QD, 5mg with best supportive care for 3 consecutive weeks, and then one week off. Tumor assessment will be performed every 4 weeks in the first 2 cycles, and every 8 weeks since the 3rd cycle, until disease progression or death. Subsequent anti-neoplastic treatment and survival status will be followed up after disease progression.
  Interventions: Drug: Fruquintinib
- Control Arm (Placebo Comparator): All subjects will receive study treatment in 4-week cycles: Placebo, QD, 5mg with best supportive care for 3 consecutive weeks, and then one week off. Tumor assessment will be performed every 4 weeks in the first 2 cycles, and every 8 weeks since the 3rd cycle, until disease progression or death. Subsequent anti-neoplastic treatment and survival status will be followed up after disease
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib is a capsule in the form of 5mg and 1mg, orally once daily. 3 weeks on/1 week off
  Other Names: HMPL-013
  Arms: Treatment Arm
Drug: Placebo — Placebo is a capsule in the form of 5mg and 1mg, orally once daily. 3 weeks on/1 week off
  Other Names: HMPL-013 placebo
  Arms: Control Arm

SUMMARY:
Fruquintinib/Placebo 5 mg, QD, orally administered under fasting conditions for 3 consecutive weeks followed by one-week off to evaluate the survival benefit of patients with advanced non-squamous NSCLC treated with Fruquintinib.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center Phase III clinical trial in patients with advanced non-squamous non-small cell lung cancer (NSCLC) treated with Fruquintinib who failed 2 lines of systemic chemotherapy or with non-tolerable toxicities.

Approximately 521 subjects will be randomized to Fruquintinib group or placebo group at a ratio of 2:1. Patients in the two groups can receive supportive treatment.

Randomization will be stratified by EGFR gene status (mutant vs. wild type) and history of treatment by VEGF inhibitors (yes vs no) .

All subjects will receive study treatment in 4-week cycles: Fruquintinib/placebo for 3 consecutive weeks, and then one week off. Tumor assessment will be performed every 4 weeks in the first 2 cycles, and every 8 weeks since the 3rd cycle, until disease progression or death. Subsequent anti-neoplastic treatment and survival status will be followed up after disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and sign the informed consent form voluntarily;
2. Histologically or cytologically diagnosed with local advanced and/or metastatic stage IIIB/IV non-squamous NSCLC;
3. Disease progressed or developed non-tolerable toxicity after 2 lines of systemic chemotherapy (not including TKI therapy); Notes: a. The first-line chemotherapy should be platinum-based doublets regimens; b. For each line of systemic therapy, at least one treatment cycle should be completed, and maintenance therapy using one of the doublets is considered as the same line of therapy; c. Previous adjuvant/neoadjuvant therapy is allowed. If disease progressed during the adjuvant/neoadjuvant therapy period or within 1 year after completion of the above treatment, it is considered that patient failed the first-line systemic chemotherapy;
4. Patients with EGFR genetic test negative; or positive with EGFR, test result but resistant or intolerable to related targeted therapies;
5. Patients with ALK test negative; or positive with ALK test result but resistant or intolerable to related targeted therapies;
6. Aged 18-75 years (inclusive);
7. Measurable disease (according to RECIST1.1);
8. ECOG Performance Status score 0-1;
9. Life expectancy >12 weeks.

Exclusion Criteria:

1. Patients who have participated in another clinical trial or received systemic anti-neoplastic therapy, radiotherapy or biotherapy within 3 weeks prior to administration of the study drug; or received EGFR-TKI treatment in the past 1 week.
2. Patients who have previously received therapy with VEGFR inhibitors;
3. Patients who have not recovered from toxicity caused by previous anti-neoplastic treatment (CTCAE > grade 1), or not completely recovered from previous surgery;
4. Patient with active brain metastasis (untreated with proper radiation therapy, showing clinical symptoms or symptom stable time less than 4 weeks, or indicated for symptomatic treatment for brain metastasis, etc.);
5. Patients with other primary malignancies within the past 5 years except basal cell carcinoma of skin or carcinoma in situ of cervix;
6. Patients with uncontrolled active infections, e.g. acute pneumonia, active hepatitis B or active hepatitis C, etc. (for patients with a history of hepatitis B, whether treated or not, HBV DNA ≥500copies or ≥ 100IU / ml);
7. Patients with dysphagia or known drug malabsorption;
8. Patients active duodenal ulcer, ulcerative colitis, intestinal obstruction and other gastrointestinal diseases or other conditions that may lead to gastrointestinal bleeding or perforation according to the investigators' judgment; or with a history of intestinal perforation or intestinal fistula;
9. Patients fulfilling any of the following criteria shall be excluded:

1) Absolute neutrophil count (ANC) <1.5×109/L, platelet <100×109/L or hemoglobin <9 g/dL within 1 week prior to enrollment;

2) Serum total bilirubin > 1.5 × upper limit of normal (ULN), alanine transaminase and aspartate aminotransferase >2.5×ULN (according to reference range in each clinical study site); ALT and AST > 5×ULN in patients with liver metastasis;

3) Clinically significant electrolyte abnormality;

4) Blood creatinine > ULN and creatinine clearance <60 ml/min;

5) Urine protein 2+ or more, or urine protein quantification ≥1.0 g/24 h;

6) Activated partial thromboplastin time (APTT) or/and INR and prothrombin time (PT) > 1.5×ULN (according to reference range in each clinical study site);

10. Patients with uncontrolled hypertension, systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg after symptomatic treatment;

11. Patients with left ventricular ejection fraction <50% (echocardiography) in heart function evaluation;

12. Patients with acute myocardial infarction, severe/unstable angina or coronary bypass surgery within 6 months prior to enrollment; cardiac insufficiency of NYHA II or above;

13. Patients who have a history of arterial thrombosis or deep venous thrombosis within 6 months prior to enrollment, history or evidence of thrombosis or bleeding tendency regardless of the severity within 2 months prior to enrollment; history of hemoptysis (i.e. coughing blood in bright red color or at least 1/2 teaspoon) within 2 weeks prior to enrollment;

14. Patients who have a history of stroke and/or transient ischemic attack within 12 months prior to enrollment;

15. Patients with skin wound, surgical site, wound site, severe mucosal ulcer or fracture without complete healing;

16. Pregnant or lactating women, or women of child bearing potential with positive pregnancy test result before the first dose;

17. Patients with child bearing potential who or whose sexual partners are not willing to take contraceptive measures;

18. Patients with any clinical or laboratory abnormalities unsuitable for participating in this clinical trial according to the investigator's judgment;

19. Patients with serious psychological or psychiatric disorders which may affect subject compliance in this clinical study;

20. Patients who are allergic to analogue of Fruquintinib and/or its inactive ingredients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | From the date of randomization until the date of death from any cause, Assessed up to 15 months
  Duration from randomization to death from any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From date of randomization until the date of first documented progression or the date of death from any cause, whichever came first, assessed up to 12 months
  Occurence of completed response or partial response after treatment, assessed by RECIST 1.1
progression free survival (PFS) | From date of randomization until the date of first documented progression or the date of death from any cause, whichever came first, assessed up to 12 months
  The duration from randomization to first documented progression or death from any cause, whichever came first, assessed by RECIST 1.1
Disease Control Rate (DCR) | From date of randomization until the date of first documented progression or the date of death from any cause, whichever came first, assessed up to 12 months
  Occurence of completed response, or partial response, or stable disease, assessed by RECIST 1.1
duration of response (DOR) | From date of randomization until the date of first documented progression or the date of death from any cause, whichever came first, assessed up to 12 months
  Duration from first documented completed response or partial response to first documented progression or death from any cause, whichever came first
safety and tolerability by incidence, severity and outcome of adverse events | From randomization to 30 days after last dose, assessed up to 13 months
  To evaluate the safety and tolerability in the two groups by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Songhua Fan, M.D., Study Director — HMP MediPharma Ltd.
Locations (11):
- China (11):
  - 307 Hospital of PLA, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Linyi Tumor Hospital, Linyi, Shandong
  - The Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - The First Affiliated Hosptial of College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided